CLINICAL TRIAL: NCT02314299
Title: A Phase 1/2, Open-Label, Dose-Escalation, Single Center, Clinical Study of MTP-131 (Ocuvia™) Topical Ophthalmic Solution in Subjects With Diabetic Macular Edema and Non-Exudative Intermediate Age-related Macular Degeneration.
Brief Title: A Study of MTP-131 Topical Ophthalmic Solution in Subjects With Diabetic Macular Edema and Non-Exudative Intermediate Age-related Macular Degeneration
Acronym: SPIOC-101
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: SPIOC-101
Record Dates: First submitted 2014-12-02; First posted 2014-12-11 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Diabetic Macular Edema; Age-related Macular Degeneration
Keywords: Macular edema; Macular degeneration; MTP-131; Ocuvia™
MeSH Terms: conditions — Macular Degeneration; Macular Edema | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Regimen (Experimental): MTP-131 (Low Dose) sterile topical ophthalmic solution twice a day into the study eye
  Interventions: Drug: MTP-131
- High Dose Regimen (Experimental): MTP-131 (High Dose) sterile topical ophthalmic solution twice a day into the study eye
  Interventions: Drug: MTP-131

INTERVENTIONS:
Drug: MTP-131

SUMMARY:
This is a Phase 1/2, open-label, dose-escalation clinical study, enrolling 21 subjects in one of the two treatment groups to determine the effects of topical ocular administration of low dose or high dose MTP-131 given twice a day in subjects with Diabetic Macular Edema and Age-Related Macular Degeneration.

ELIGIBILITY:
Inclusion Criteria:

* General:

  1. Adults aged ≥18 and ≤ 80 years
  2. Women of childbearing potential must have a negative urine pregnancy test at Baseline and agree to use a highly effective method of contraception throughout the study and 60 days after the last dose of study drug.
* DME Treatment Group:

  1. Central subfield thickness (CST) ≥325 microns as measured by spectral domain optical coherence tomography (SD-OCT) at Screening and Baseline Visits
  2. BCVA (ETDRS) no better than 20/25 in the study eye
  3. BCVA (ETDRS) no worse than 20/640 in either eye
* AMD Treatment Group:

  1. Non-exudative, intermediate age-related macular degeneration defined as an eye(s) having extensive intermediate drusen (10 or more drusen 63μm - 124μm) or large drusen (1 or more ≥125 μm) with no evidence of advanced AMD (i.e., no choroidal neovascularization or macular atrophy)
  2. BCVA (ETDRS) no worse than 20/400 in either eye

Exclusion Criteria:

* General:

  1. Inability to self-administer eye drops
  2. Current use of or likely need for systemic medications known to be toxic to the lens, retina or optic nerve (for example deferoxamine, chloroquine/hydroxychloroquine [Plaquenil], tamoxifen, phenothiazines and ethambutol)
  3. Any medical condition that, in the opinion of the investigator, would preclude safe participation in the study or completion of all study requirements and examinations
  4. Have a glycosylated hemoglobin (HbA1c) ≥ 12%
* Ocular Conditions:

  1. Any ocular condition in the study eye that in the opinion of the investigator would prevent improvement in visual acuity or successful completion of any study examination
  2. Ocular hypertension or glaucoma, dry eye, and any other ocular pathology in the study eye requiring treatment with topical ophthalmic drops

     * Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of systemic and ocular adverse events | From Baseline to Day 28
Change from Baseline in vital sign measurements | From Baseline to Day 28
Change from Baseline in best corrected visual acuity (BCVA) as measured with the early treatment diabetic retinopathy study (ETDRS) scale | From Baseline to Day 28
Change from Baseline in slit lamp examinations | From Baseline to Day 28
Change from Baseline in intraocular pressure | From Baseline to Day 28
Change from Baseline in dilated fundoscopic examinations | From Baseline to Day 28
Change from Baseline in central subfield thickness | From Baseline to Day 28

SECONDARY OUTCOMES:
Change in central subfield thickness | From Baseline to Day 28
  Diabetic Macular Edema (DME) subjects only
Change from Baseline in widefield angiography | From Baseline to Day 28
  Diabetic Macular Edema (DME) subjects only
Change from Baseline in fundus autofluorescence pattern including the occurrence of and aggregate size of areas of macular atrophy | From Baseline to Day 28
  Age-Related Macular Degeneration (AMD) subjects only
Change from Baseline in best corrected visual acuity (BCVA) as measured with the early treatment diabetic retinopathy study (ETDRS) scale | From baseline to Day 28
  All subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Boston, Massachusetts, United States